CLINICAL TRIAL: NCT06167174
Title: Exploring Biomarkers for Therapeutic Response of Lupus Nephritis Based on Multi Omics
Brief Title: Exploring Biomarkers for Therapeutic Response of Lupus Nephritis Based on Multi Omics Analysis
Status: Recruiting | Type: Observational
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CSTAR-K2939
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood, kidney tissues and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMF treatment: Patients that have been diagnosed as III/IV ± V LN and treated with MMF 2g/d in combination with glucocorticoid.
- CYC treatment: Patients that have been diagnosed as III/IV ± V LN and treated with CYC 0.5g IV per two weeks in combination with glucocorticoid.

SUMMARY:
This is an observational study of patients with lupus nephritis aiming to find biomarkers that can predict patients' response to immunosuppressants. We planed to collect 100 lupus nephritis patients' peripheral blood,kidney tissues and urine before and after treatment (mycophenolate mofetil or cyclophosphamide, in combination with glucocorticoids). Then multi omics analysis, including single cell RNA-seq, ATAC-seq and CITE-seq, will be performed to find new biomarkers for patients' response and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16-60 years.
2. Fulfilling the 2012 SLICC classification for SLE.
3. Renal biopsy pathology was clearly classified as III \ IV \ V+III \ V+IV within 6 months.
4. Renal biopsy reveals active disease.
5. 24-hour urinary protein was tested twice within two weeks, both of which were greater than 1g.
6. The patients have never received glucocorticoid/immunosuppressants or received standard treatment for more than 1 month without change. The standard treatment should fulfill: a. prednisone 0-20mg/day, or equivalent other glucocorticoids; b. acceptable immunosuppressants, including Tacrolimus ≤ 4mg/d, methotrexate ≤ 15mg/week, azathioprine ≤ 100mg/d and MMF ≤ 1g/d.
7. Informed consent obtained.

Exclusion Criteria:

1. Other concomitant connective tissue diseases or autoimmune diseases.
2. Neuropsychiatric lupus, alveolar hemorrhage, retinal lesions, pulmonary arterial hypertension, or other severe organ involvement.
3. Pregnant or lactating women.
4. Current infections that require antibiotic or antiviral treatment.
5. Other kidney diseases.
6. Platelet < 50×10^9/L.
7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) that is greater than 1.5 times the upper limit of the normal value.
8. Total bilirubin or blood lipid that is greater than 2 times the upper limit of the normal value.
9. Other conditions that not suitable for inclusion in the study, assessed by the investigators.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients visit Rheumatology and Immunology Department of Peking Union Medical College Hospital and fulfill the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-05 (Estimated); Primary Completion 2027-12-05 (Estimated); Study Completion 2028-12-05 (Estimated)

PRIMARY OUTCOMES:
Treatment response of patients | 24 weeks
  The proportion of patients who achieve complete response, partial response or no response 24 weeks after baseline

SECONDARY OUTCOMES:
Disease progression | 24 weeks
  Clinical indices that can indicate the progression of disease, including 24-hour urinary protein, routine urine and blood tests, immune indices and patients' syndromes, will be evaluated at 4, 12, 24 weeks after baseline to monitor the progression of lupus nephritis.
Adverse events during the study | 24 weeks
  All adverse events, severe adverse events and proportion of patients who discontinued the treatment due to adverse events within the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Xinping Tian, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No